CLINICAL TRIAL: NCT05643105
Title: Prospective Observational Multicenter Study of Anastomotic Leakage After Colon Cancer Surgery (ANACO II).
Brief Title: Anastomotic Leakage After Colon Cancer Surgery
Acronym: ANACO II
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Spanish Association of Surgeons (AEC) (Other); Hospital Universitario La Fe (Other); Complejo Hospitalario Universitario de Vigo (Other)
Responsible Party: Principal Investigator, Carlos Cerdán Santacruz, Consultant. Colorectal Surgery Department. Principal Investigator, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Other Study IDs: 10/22-4851
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Adult Patients; Intestinal Continuity (Anastomosis); Colon Cancer
Keywords: colon cancer; anastomotic leakage
MeSH Terms: conditions — Colonic Neoplasms; Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colon cancer patients with intestinal anastomosis: There is a single cohort of patients, the one operated on for colon cancer with intestinal continuity construction through an anastomosis without derivative stoma construction of any kind.
  Interventions: Procedure: Any kind of colectomy

INTERVENTIONS:
Procedure: Any kind of colectomy — This is a registry of surgical patients with colon cancer that are managed following current clinical practice in each participating center. The aim of this research is studying anastomotic leak rates and posible risk factors.
  Other Names: Adjuvant chemotherapy when necessary following current clinical practice

SUMMARY:
Anastomotic leak (AL) is one of the most feared complications after colon cancer (CC) surgery. The incidence varies according to the studies, the definition used and the location of the excised segment.

In some of the series described, AL incidence have hardly changed, despite the evolution of the technique and technological improvements. The leak rate obtained in the only Spanish prospective multicenter observational study at national level was 9% (ANACO study).

The aim of the present study is to determine the current rate of AL in our country, 10 years after the ANACO study, to determine if there has been any evolution and to analyze the factors associated with it. For this purpose, AL is defined with the same criteria as in the first study, as leakage of luminal contents through the junction between two hollow visceras, diagnosed radiologically (radiography with soluble enema or CT with collection adjacent to the anastomosis), clinically (extravasation of luminal contents or gas through the wound or drainage), endoscopically or intraoperatively. To compare AL rates throughout this decade, a 60-day follow-up will be performed, the same as in the ANACO study.

As a modification respect to the ANACO study protocol, the aim is to analyze the possible influence of AL and perioperative intra-abdominal infection on short-term oncologic prognosis, with a one-year follow-up. This question has hardly been studied in prospective multicenter studies to date.

The variables to be collected are divided into demographic (information about the hospital center, patient comorbidities), diagnostic variables (analytical values, diagnostic reason, neoadjuvant, localization, TNM), surgical variables (type of surgery, preparation, intention, intraoperative findings and complications, type of resection and anastomosis), admission (AL, other complications), histology, 60-day follow-up (AL, readmissions), one-year follow-up (readmissions, local recurrence, peritoneal and distant recurrence).

Patients included in the study must be >18 years old undergoing oncologic surgery for CC located 15 cm above the anal margin, with preoperative histological confirmation or with endoscopic suspicion of infiltrating lesion or with radiological suspicion in the context of urgent surgery. Intestinal continuity (anastomosis) should be reconstructed and a derivative stoma should not be associated in the same surgery. According to ANACO data and follow-up times according to the primary objective (AL) at 60 days and the secondary objective (oncologic prognosis) with annual follow-up, inclusion will be carried out until the 1628 individuals required according to the sample size calculation performed are included.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old undergoing oncologic surgery for CC located 15 cm above the anal margin, with preoperative histological confirmation or with endoscopic suspicion of infiltrating lesion or with radiological suspicion in the context of urgent surgery. Intestinal continuity (anastomosis) should be reconstructed in the same surgery.

Exclusion Criteria:

* Derivative stoma in the same surgery
* Palliative surgery
* Definitive stoma creation without anastomosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologic surgery for colon cancer located 15 cm above the anal margin, with preoperative histological confirmation or with endoscopic suspicion of infiltrating lesion or with radiological suspicion in the context of urgent surgery
Sampling Method: Non-Probability Sample
Enrollment: 1628 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | 60 days

SECONDARY OUTCOMES:
Overall postoperative complications | 60 days
Local recurrence | 1 year

OTHER OUTCOMES:
Minimally invasive surgery use | 1 day
  Amount of patients that are operated on for colon cancer using minimally invasive approaches, both laparoscopic or robotic
Intraoperative complications | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Cerdán, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Carlos Cerdán Santacruz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
It is the intention of the authors to share data collected through an official data repository such as Mendeley, for example.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From three months after recruitment after 3 months of follow-up ending.
Access Criteria: Under demand.